CLINICAL TRIAL: NCT00666341
Title: A Double-blind Placebo-controlled Dose-response Study for Evaluation of Safety and Efficacy of Immunotherapy With a Cocktail of Recombinant Major Allergens of Timothy Grass Pollen (Phleum Pratense) Adsorbed to Aluminium Hydroxide in Patients With IgE-mediated Allergic Rhinitis/Rhinoconjunctivitis With or Without Bronchial Asthma
Brief Title: Dose-Response-Study With a Recombinant Cocktail of Phleum (rPhleum) Allergens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AL0701rP; 2007-002808-18 (EudraCT Number)
Record Dates: First submitted 2008-04-21; First posted 2008-04-24 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Type I-Allergy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo: Al(OH)3-Placebos with histamine-dihydrochloride analogue Allergen-Adsorbate rPhleum strengthes 1 to 4.
  Interventions: Drug: placebo
- 20 μg rPhleum Immunotherapy (Experimental): Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 1 (20 μg)
  Interventions: Biological: rPhleum
- 40 μg rPhleum Immunotherapy (Experimental): Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 2 (40 μg)
  Interventions: Biological: rPhleum
- 80 μg rPhleum Immunotherapy (Experimental): Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 3 (80 μg)
  Interventions: Biological: rPhleum
- 120 μg rPhleum Immunotherapy (Experimental): Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 4 (120 μg)
  Interventions: Biological: rPhleum

INTERVENTIONS:
Drug: placebo — Placebo: Al(OH)3-Placebos with histamine-dihydrochloride analogue Allergen-Adsorbate rPhleum strengthes 1 to 4.
  Other Names: Comparator
  Arms: Placebo
Biological: rPhleum — Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 1 (20 μg)
  Other Names: Specific Immunotherapy
  Arms: 20 μg rPhleum Immunotherapy
Biological: rPhleum — Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 2 (40 μg)
  Other Names: Specific Immunotherapy
  Arms: 40 μg rPhleum Immunotherapy
Biological: rPhleum — Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 3 (80 μg)
  Other Names: Specific Immunotherapy
  Arms: 80 μg rPhleum Immunotherapy
Biological: rPhleum — Cocktail of recombinant major allergens of Phleum pratense (timothy grass) with strength 4 (120 μg)
  Other Names: Specific Immunotherapy
  Arms: 120 μg rPhleum Immunotherapy

SUMMARY:
Dose-response trial with a cocktail of recombinant major allergens of Timothy Grass Pollen (Phleum pratense)

ELIGIBILITY:
Inclusion Criteria:

* main symptoms of allergic rhinitis/rhinoconjunctivitis with or without controlled asthma against grass pollen allergens
* positive SPT
* positive EAST
* positive specific provocation test

Exclusion Criteria:

* serious chronic diseases
* other perennial allergies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Systemic reaction (according to Tryba) | uptitration phase
  Number of patients with at least one systemic reaction (according to Tryba Grade 1-4) with possible, probable or definite relationship to the study medication determined at the end of the uptitration phase.

SECONDARY OUTCOMES:
Late Phase Reactions | before and at the end of the double-blind phase
  Changes of the Late Phase Reactions in specific intracutaneous test with natural allergen before and at the end of the double-blind placebo controlled phase before grass pollen season.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Hörmann, MD, Study Chair — Universitätsklinikum Mannheim GMBH
Locations (1):
- Prof. Dr. med. Ludger Klimek, Wiesbaden, Baden-W., Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-002808-18/DE